CLINICAL TRIAL: NCT05866822
Title: Adapted Physical Activity Education in Patients With Neurocognitive Disorder: Single-blind, Single-center Randomized Controlled Trial
Brief Title: Adapted Physical Activity Education in Patients With Neurocognitive Disorder
Acronym: EduAPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-AOI-10
Record Dates: First submitted 2023-04-28; First posted 2023-05-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APA (adapted physical activity) (Active Comparator): 24 APA sessions will take place, there will be 2 sessions a week for 12 weeks which will include global exercises for the upper and lower limb. One session will be 1 hour long and supervised by professionals. It will be divided in 4 cycles which will be differentiated by the intensity of its components: aerobic, strength, speed, balance, coordination and flexibility. The intensity of the sessions will be measured by RPE and heart rate monitor,
  Interventions: Other: APA
- APA (adapted physical activity) + physical activity education (PAE) (Experimental): 24 APA sessions will take place, there will be 2 sessions a week for 12 weeks which will include global exercises for the upper and lower limb. One session will be 1 hour long and supervised by professionals. It will be divided in 4 cycles which will be differentiated by the intensity of its components: aerobic, strength, speed, balance, coordination and flexibility. The intensity of the sessions will be measured by RPE and heart rate monitor,
  + 8 individuals sessions of PAE (one per week, half an hour long) that will consist of advising and setting weekly goals related to improving PA level and sedentary behavior
  Interventions: Other: APA; Other: PAE

INTERVENTIONS:
Other: APA — 24 APA sessions
Other: PAE — 8 individuals sessions of PAE
  Arms: APA (adapted physical activity) + physical activity education (PAE)

SUMMARY:
This study aims to compare the effect of a program of Adapted Physical Activity (APA) versus the same program combined with a physical activity education program (PAE). Patients suffering from neurocognitive disorders (mild or early major) will be randomized into one of the two conditions. 3 complete evaluations will be done (inclusion M0, after 3 month of intervention M3, 3 months after the end of the intervention M6). The team except that APA+PEA will be more effectiv than the APA solely, on the following criteria : level of physical activity, cogntive function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* mild neurocognitive disorder or early major neurocognitive disorder

Exclusion Criteria:

* Medical pathology involving the vital prognosis in the short term
* Major neurocognitive disorder at moderate stage and beyond (DSM 5) and/or MMSE < 20
* Unbalanced depressive syndrom
* Contraindication to the practice of the exercises proposed during the study;
* Major hearing or visual impairment;
* Sufficiently active with regard to the daily recommendations described by the WHO

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
physical activity level | at inclusion
  evolution of physical activity level will be assessed by actimetry on a 7 days period mesured by IPAQ score
physical activity level | at 3 months after inclusion
  evolution of physical activity level will be assessed by actimetry on a 7 days period mesured by IPAQ score
physical activity level | at 6 months after inclusion
  evolution of physical activity level will be assessed by actimetry on a 7 days period mesured by IPAQ score

SECONDARY OUTCOMES:
global cognition | at inclusion
  global cognition will be assessed by a MMSE test (Mini Mental State Examination) mesured by a score
global cognition | at 3 months after inclusion
  global cognition will be assessed by a MMSE test (Mini Mental State Examination) mesured by a score
global cognition | at 6 months after inclusion
  global cognition will be assessed by a MMSE test (Mini Mental State Examination) mesured by a score
executive functions | at inclusion
  executiv functions will be assessed by FAB (frontal assessment battery)
executive functions | at 3 months after inclusion
  executiv functions will be assessed by FAB (frontal assessment battery)
executive functions | at 6 months after inclusion
  executiv functions will be assessed by FAB (frontal assessment battery)
executive functions (FAB) | at inclusion
  executiv functions will be assessed by FAB (frontal assessment battery) giving a score
executive functions (FAB) | at 3 months after inclusion
  executiv functions will be assessed by FAB (frontal assessment battery) giving a score
executive functions (FAB) | at 6 months after inclusion
  executiv functions will be assessed by FAB (frontal assessment battery) giving a score
executive functions (TMT) | at inclusion
  executiv functions will be assessed by TMT (frontal assessment battery) - giving a score
executive functions (TMT) | at 3 months after inclusion
  executiv functions will be assessed by TMT (frontal assessment battery) - giving a score
executive functions (TMT) | at 6 months after inclusion
  executiv functions will be assessed by TMT (frontal assessment battery) - giving a score
cardiovascular performance | at inclusion
  Cardiovascular performance will be evaluated through a effort test that will be performed on a stationary bicycle ergometer connected to a portable gas exchange analysis system in ml/kg/min
cardiovascular performance | at 3 months after inclusion
  Cardiovascular performance will be evaluated through a effort test that will be performed on a stationary bicycle ergometer connected to a portable gas exchange analysis system in ml/kg/min
cardiovascular performance | at 6 months after inclusion
  Cardiovascular performance will be evaluated through a effort test that will be performed on a stationary bicycle ergometer connected to a portable gas exchange analysis system in ml/kg/min
power - physical condition | at inclusion
  physical condition will be asessed by lower extremity power (isokinetic ergometer) with a score
power - physical condition | at 3 months after inclusion
  physical condition will be asessed by lower extremity power (isokinetic ergometer) with a score
power - physical condition | at 6 months after inclusion
  physical condition will be asessed by lower extremity power (isokinetic ergometer) with a score
strenght - physical condition | at inclusion
  physical condition will be asessed by grip strength (hand grip) with a score
strenght - physical condition | at 3 months after inclusion
  physical condition will be asessed by grip strength (hand grip) with a score
strenght - physical condition | at 6 months after inclusion
  physical condition will be asessed by grip strength (hand grip) with a score
evaluation of quality of life | at inclusion
  quality of life will be assessed by SF 12 a short version of the MEDICAL OUTCOME STUDY SHORT FORME GENERAL HEALTH SURVEY (score)
evaluation of quality of life | at 3 months after inclusion
  quality of life will be assessed by SF 12 a short version of the MEDICAL OUTCOME STUDY SHORT FORME GENERAL HEALTH SURVEY (score)
evaluation of quality of life | at 6 months after inclusion
  quality of life will be assessed by SF 12 a short version of the MEDICAL OUTCOME STUDY SHORT FORME GENERAL HEALTH SURVEY (score)
anxiety and depression | at inclusion
  anxiety and depression will be assessed by the HADS " Hospital Anxiety and Depression Scale " and giving a score
anxiety and depression | at 3 months after inclusion
  anxiety and depression will be assessed by the HADS " Hospital Anxiety and Depression Scale " and giving a score
anxiety and depression | at 6 months after inclusion
  anxiety and depression will be assessed by the HADS " Hospital Anxiety and Depression Scale " and giving a score
apathy | at inclusion
  apathy will be assessed by the apathy inventory questionnary and givig a score
apathy | at 3 months after inclusion
  apathy will be assessed by the apathy inventory questionnary and givig a score
apathy | at 6 months after inclusion
  apathy will be assessed by the apathy inventory questionnary and givig a score

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France